CLINICAL TRIAL: NCT06000228
Title: "Effect of Vestibular Depth on Root Coverage Predictability in Miller Class III/Recession Type 2 Labial Gingival Recession Treated With Minimally Invasive Technique Using Connective Tissue Graft: A Prospective Cohort Study
Brief Title: Effect of Vestibular Depth on Predictability of Miller Class III/ RT2 Gingival Recession Coverage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sushma Periodontics 2022
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shallow vestibule (Experimental): Miller class III/ RT2 labial gingival recession associated with vestibular depth less than 6mm
  Interventions: Procedure: Recession coverage with CTG using minimally invasive access technique in shallow vestibule
- Deep vestibule (Active Comparator): Miller class III/ RT2 labial gingival recession associated with vestibular depth more than 6mm
  Interventions: Procedure: Recession coverage with CTG using minimally invasive access technique in deep vestibule

INTERVENTIONS:
Procedure: Recession coverage with CTG using minimally invasive access technique in shallow vestibule — After enrolment, participants will be instructed about oral hygiene and undergo nonsurgical periodontal treatment in the form of scaling and root planing using ultrasonic and hand instruments as needed. After resolution of inflammation, a full thickness tunnel will be preapred using minimally invasive access technique under local anesthesia with the aid of specific tunnelling instruments and connective tissue graft will be procured from the palate or tuberosity area for root coverage procedure by single incision technique.
  Arms: Shallow vestibule
Procedure: Recession coverage with CTG using minimally invasive access technique in deep vestibule — After enrolment, participants will be instructed about oral hygiene and undergo nonsurgical periodontal treatment in the form of scaling and root planing using ultrasonic and hand instruments as needed. After resolution of inflammation, a full thickness tunnel will be preapred using minimally invasive access technique under local anesthesia with the aid of specific tunnelling instruments and connective tissue graft will be procured from the palate or tuberosity area for root coverage procedure by single incision technique.
  Arms: Deep vestibule

SUMMARY:
Aim of this study is to assess the influence of vestibular depth on root coverage in Miller class III/ Cairo RT2 gingival recession when treated with minimally invasive technique using connective tissue graft.

DETAILED DESCRIPTION:
Gingival recession is defined as partial exposure of the root surface to the oral cavity because of apical migration of the gingival margin (GM) with respect to the cemento-enamel junction (CEJ). Miller class III/Cairo RT2 gingival recession most common gingival recession where patient complaint of root sensitivity, root caries and wedge shape defect. Several mucogingival approaches have been proposed such as tunnel techniques, coronally advanced flap(most common), connective tissue graft, rotated flap. Local factor that influences the surgical intervention and outcome therapy is interproximal bone and attachment level, marginal gingival thickness (MGT), width of attached gingiva, and recession defect depth (RD) clinical attachment level (CAL). In recent publication Aroca et al. studied influence of distance from tip of the papilla and the contact point (DCP) on recession coverage outcome and concluded that the probability to obtain a complete root coverage decreases when the DCP at baseline increases. Another finding of recent case series shown association of vestibular depth (VD) and outcome in terms of % root coverage (%RC) and complete complete coverage (CRC) and revealed that each additional 1mm VD increased 2.75 times the probability of achieving CRC but they have not compared the root coverage outcome in deep and shallow vestibular depth. Therefore, this study will be conducted in Miller class III/RT2 labial gingival recession to observed the impact of vestibular depth on root coverage when treating with minimally invasive technique using connective tissue graft.

AIM AND OBJECTIVE To assess the influence of vestibular depth on root coverage in Miller class III/ Cairo RT2 gingival recession when treated with minimally invasive technique using connective tissue graft.

Primary objective Comparative evaluation of percentage of recession coverage and complete root coverage in shallow and deep vestibular depth in Miller class III/ Cairo RT2 when treated with minimally invasive technique using connective tissue graft and also evaluated RD, RW, Gingiva phenotype, patient-based evaluation of pain and hypersensitivity by visual analogue scale(VAS)

Secondary objective To assess the improvement to other clinical parameter which will include clinical attachment level (CAL), Interdental clinical attachment, Mid buccal clinical attachment, Pocket probing depth (PPD), Bleeding on probing (BOP), Plaque index (PI), Gingival thickness (GT), Keratinized tissue width (KTW), Root aesthetic score (RES).

STUDY DESIGN Prospective cohort study

STUDY SETTING Hospital based study, and will be conducted in department of Periodontics, Post graduate institute of dental science, Rohtak.

STUDY PERIOD 12 to 14 months follow up

STUDY SUBJECT Systemically healthy individuals with Miller class III/Cairo RT2 labial gingival recession will be recruited from the outpatient department of periodontology.

Patients fulfilling the eligibility criteria will be enrolled in the study after obtaining an informed written consent.

MATERIAL AND METHOD

Patient will be educated about the procedure and its implication. Scaling and root planing is performed and then participants will be instructed about oral hygiene and undergo intervention therapy.

After administration of local anesthesia, exposed root surface will be planed using curettes or by using bur to reduce the prominent root. With a minimally invasive access technique a full thickness tunnel will be prepared with specific tunneling instruments, extending it sufficiently beyond the mucogingival line into alveolar mucosa, this will be done to completely releasing the tunnel-papillae complex, thus facilitating its passive coronal replacement. connective tissue graft will be procured from the palate or tuberosity area for root coverage procedure by single incision technique. The palatal wound will be sutured (5-0) to obtain primary wound closure Then after surgery patient will be recalled after 10 -12 days and then again at 1, 3, 6 months.

STUDY GROUPS

Experimental group- Miller class III/RT2 labial gingival recession associated with shallow vestibule.

Active comparator- Miller class III/RT2 labial gingival recession associated with deep vestibule.

STATISTICAL ANALYSIS Data recorded will be processed by standard statistical analysis. The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to distribution of data. If it is in normal distribution inter group comparison will be done by using Independent T test and paired t test will be used for intragroup comparison and if non-normal distribution of data, inter group comparison will be done by Mann-Whitney U test and intragroup by signed rank test. The Chi square test will be applied to analysed categoric data. Correlation and association between predictors and dependent variables will be analysed by correlation analysis and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years) presenting with isolated Miller class III / Cairo RT2 labial gingival recession defect with deep and shallow vestibular defect.
2. Absence of clinical tooth mobility.
3. Age >18 years old.
4. A full mouth plaque index and full mouth bleeding index < 20%
5. Patient showing adequate compliance and willing to participate in the study.
6. CAL (clinical attachment level), RD (recession depth) and KTW (keratinized tissue depth) will be comparable and matched in both the groups.

Exclusion Criteria:

(1) full-mouth plaque and bleeding score >20%; (2) non smoker; (3) systemic contraindications for periodontal surgery; (4) taking medications known to affect gingival homeostasis or interfere with wound healing; (5) pregnancy; (6) active orthodontic therapy; (7) previous periodontal surgery, caries, or restorations in the experimental site(s); and (8) malpositioned /crowded teeth.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
percentage root coverage | 12-14 months
  percentage of root coverage is calculated using formula: Preoperative recession depth-postoperative recession depth/ preoperative recession depth × 100

CONTACTS AND LOCATIONS:
Overall Officials: sushma Kumari, BDS, Principal Investigator — Postgraduate Institute of Dental Sciences Rohtak
Locations (1):
- Shikha Tewari, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No